CLINICAL TRIAL: NCT03426956
Title: Impact of Canaglifloxin on Gut Hormone Secretion After Gastric Bypass
Brief Title: Glucose Absorption and Gut Hormone Secretion After Gastric Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christoffer Martinussen, Principal investigator, Medical Doctor, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CM-CANA-18
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Overweight
Keywords: Glucagon-like Peptide-1; Glucose; Gastric bypass; Bariatric surgery; Obesity; Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus | interventions — Glucose; Canagliflozin

STUDY DESIGN:
Intervention Model Description: 10 gastric bypass patients
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose (Experimental)
  Interventions: Dietary Supplement: Glucose
- Glucose + Canagliflozin (Experimental)
  Interventions: Dietary Supplement: Glucose + Canagliflozin

INTERVENTIONS:
Dietary Supplement: Glucose — Ingestion of glucose (50 g) dissolved in 200 ml water.
  Arms: Glucose
Dietary Supplement: Glucose + Canagliflozin — Ingestion of glucose (50 g) dissolved in 200 ml water combined with the SGLT-1/SGLT-2 inhibitor canagliflozin.
  Arms: Glucose + Canagliflozin

SUMMARY:
To investigate the impact of canagliflozin on secretion of gut hormones, in particular glucagon-like peptide 1 (GLP-1) in gastric bypass operated patients.

DETAILED DESCRIPTION:
Glucose is a potent stimulus for GLP-1 secretion after gastric bypass surgery and the SGLT-1 transporter appears to be crucial for this response. The study will investigate the effects of SGLT-1/SGLT-2 inhibition (by canagliflozin) on secretion of GLP-1 and other gut hormones after gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

•Uncomplicated gastric bypass surgery performed minimum 12 months prior to study

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus prior to or after gastric bypass surgery
* Pregnancy or breastfeeding
* Haemoglobin levels below 6,5 mM

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-02-08 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference in GLP-1 secretion (evaluated by iAUC). | 0-240 min following glucose ingestion
  Comparison of the GLP-1 responses (evaluated by iAUC) between the two test days.

SECONDARY OUTCOMES:
Difference in glucose responses between the two test days. | 0-240 min following glucose ingestion
Difference in insulin responses between the two test days. | 0-240 min following glucose ingestion
Difference in C-peptide responses between the two test days. | 0-240 min following glucose ingestion
Difference in Gastric Inhibitory Peptide (GIP) responses (evaluated by iAUC) between the two test days. | 0-240 min following glucose ingestion
Difference in peptide YY (PYY) responses (evaluated by iAUC) between the two test days. | 0-240 min following carbohydrate ingestion
Difference in glucagon responses (evaluated by iAUC) between the two test days. | 0-240 min following glucose ingestion
Difference in oxyntomodulin responses (evaluated by iAUC) between the two test days. | 0-240 min following carbohydrate ingestion
Difference in cholecystokinin (CCK) responses (evaluated by iAUC) between the two test days. | 0-240 min following glucose ingestion
Difference in bile acid responses (evaluated by iAUC) between the two test days. | 0-240 min following glucose ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Endocrinology, Hvidovre, Denmark